CLINICAL TRIAL: NCT05352269
Title: Safety and Tolerability of Xbiome Gut Microbial Capsule XBI-302 in Healthy Volunteers
Brief Title: Safety and Tolerability of FMT Capsules in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Xbiome Biotech Co., Ltd. (Industry)
Collaborators: Beijing Improve-Quality Tech.Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: XBI302CT9001
Record Dates: First submitted 2022-04-12; First posted 2022-04-28 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Acute-graft-versus-host Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 XBI-302 (Experimental): 40 XBI-302 capsules in 1 day
  Interventions: Biological: XBI-302
- Cohort 1 Placebo (Placebo Comparator): 40 placebo capsules in 1 day
  Interventions: Biological: XBI-302 Placebo
- Cohort 2 XBI-302 (Experimental): 80 XBI-302 capsules over 2 days
  Interventions: Biological: XBI-302
- Cohort 2 Placebo (Placebo Comparator): 80 placebo capsules over 2 days
  Interventions: Biological: XBI-302 Placebo
- Cohort 3 XBI-302 (Experimental): 40 XBI-302 capsules per day, once a week for 4 weeks.
  Interventions: Biological: XBI-302
- Cohort 3 Placebo (Placebo Comparator): 40 placebo capsules per day, once a week for 4 weeks.
  Interventions: Biological: XBI-302 Placebo
- Cohort 4 XBI-302 (Experimental): 80 XBI-302 capsules over 2 days, once a week for 4 weeks.
  Interventions: Biological: XBI-302
- Cohort 4 Placebo (Placebo Comparator): 80 placebo capsules over 2 days, once a week for 4 weeks.
  Interventions: Biological: XBI-302 Placebo

INTERVENTIONS:
Biological: XBI-302 — Fecal Microbiota Transplantation Capsules
  Arms: Cohort 1 XBI-302; Cohort 2 XBI-302; Cohort 3 XBI-302; Cohort 4 XBI-302
Biological: XBI-302 Placebo — XBI-302 Placebo
  Arms: Cohort 1 Placebo; Cohort 2 Placebo; Cohort 3 Placebo; Cohort 4 Placebo

SUMMARY:
This is a two-part, randomized, double-blind, placebo-controlled, single center study to investigate the safety and tolerability of XBI-302 administered orally in healthy volunteers. The hypothesis of this study is that XBI-302 is safe and well tolerated with the proposed dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate and sign the ICF.
2. Healthy adults 18-55 years of age, male and female.
3. For women of childbearing age, negative serum pregnancy test at Screening and negative serum pregnancy test confirmed at the admission to the Phase 1 unit.
4. Female participants must not be pregnant, lactating, or actively trying to become pregnant. Participants who are premenopausal and of childbearing potential must have two negative pregnancy tests (serum) and both female and male participants must use medically acceptable and effective contraceptive methods during the study period, including:

   1. Having a male partner who is sterile prior to the female participant's entry into the study and is the sole sexual partner for that female participant
   2. Use of double-barrier methods of contraception; condoms with the use of caps (with spermicide) and intra-uterine devices are acceptable
   3. True abstinence, when this is in line with the preferred and usual lifestyle of the participant (Note: period abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
5. Clinical laboratory test values (hematology, blood chemistry, routine stool test, urinalysis, etc.) are in the normal ranges or although it was outside the normal limits, the researchers determined that the participant will still be eligible within the screening period.
6. Participants have a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m2) inclusive, and a body weight of at least 45 kilograms (kg).

Exclusion Criteria:

1. History of cardiovascular disease, immune system disease, malignant disease such as cancer, nervous system disease, hematological disease, endocrinological disease, and/or any other diseases that in the opinion of the investigator could impact assessments of safety or the gut microbiome.
2. Significant past medical history of GI conditions including inflammatory bowel disease, irritable bowel syndrome, celiac disease, history of GI malignancy or polyposis, C. difficile infection in past year.
3. GI symptoms that occur more than four times a month including acid reflux, nausea, vomiting, diarrhea, abdominal pain or cramps, abdominal distension, bloating, constipation.
4. Used oral antibiotics within 4 weeks prior to the first FMT dosing.
5. HIV infection and/or HBV/HCV infection.
6. Active tuberculosis and undergoing treatment.
7. History of mental illness, drug or alcohol abuse and/or any other behavioral issues that may impact study compliance.
8. Lactating women or participants who plan to become pregnant or conceive within half a year.
9. History of severe hypersensitivity (may cause difficulty in breathing).
10. Alcohol breathalyzer test positive, urine drug screening test positive, and/or smoker.
11. Participated in any other clinical trials within 3 months of first dose.
12. Participants with history of bowel or gastrointestinal surgery.
13. Participants who are immunosuppressed or immunocompromised, either by genetic, acquired or secondary to medication.
14. Participants who are experiencing symptoms associated with COVID-19 (including but not limited to cough, fever, shortness of breath, nausea, diarrhea, anhedonia, anosmia, ageusia or severe fatigue).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of all AEs and SAEs | Day 28
  The incidence and severity of all AEs and SAEs that are determined to be related to XBI-302 through Day 28.

SECONDARY OUTCOMES:
The incidence of all AEs and SAEs | Day 28 and Week 12
  The incidence of all AEs and SAEs through Day 28 and Week 12.
Change in laboratory data of pre- and post-intervention as a measure of safety. | Baseline, Weeks 1, 2, 3, 4, and 12 (if applicable for the arm)
  Compare changes laboratory data via hematology, blood chemistry, urinalysis, and routine stool testing before and after using FMT capsules.
Change in functions of all organ systems via standard complete physical examinations. | Baseline, Weeks 1, 2, 3, 4, and 12 (if applicable for the arm)
  Change in functions of all organ systems via standard complete physical examinations.
Change in functions of heart, lungs, abdomen and other organ that involve the gastrointestinal tract and digestive system via targeted physical examinations. | Baseline, Weeks 1, 2, 3, 4, and 12 (if applicable for the arm)
  Change in functions of heart, lungs, abdomen and other organ that involve the gastrointestinal tract and digestive system via targeted physical examinations.
Change in vital signs in ear temperature, pulse, respirations, and blood pressure as a measure of safety. | Baseline, Weeks 1, 2, 3, 4, and 12 (if applicable for the arm)
  Change in vital signs in ear temperature, pulse, respirations, and blood pressure as a measure of safety.
The incidence of gastrointestinal AEs | Weeks 1, 2, 3, and 4 (if applicable for the arm)
  Compare the incidence of gastrointestinal AEs on the dosing day(s) between treatment groups.
The level of difficulty of swallowing FMT capsules as a measure of tolerability. | Weeks 1, 2, 3, and 4 (if applicable for the arm)
  Estimate degree of difficulty of swallowing FMT capsules via daily diary cards by selecting easy, ok, hard (must rest frequently to complete all capsules), or very hard (stuck to my throat all the time, took a long time to finish all capsules).
The subjective experience of the taste acceptance as a measure of tolerability. | Weeks 1, 2, 3, and 4 (if applicable for the arm)
  Estimate degree of taste acceptance of FMT capsules via daily diary cards by selecting none, ok, a strange taste, or strong taste that makes me nauseous.
The gut microbiome profile | Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, and 12 (if applicable for the arm)
  Compare the gut microbiome profile before and after the transplantation between treatment groups.
The gut microbiome profile | Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, and 12 (if applicable for the arm)
  Compare the gut microbiome profile before and after the transplantation between donors and participants.
The colonization of microbiota from donor | Baseline, Weeks 1, 2, 3, 4, 6, 8, 10, and 12 (if applicable for the arm)
  Compare the effects of diet and lifestyle on the colonization of microbiota from donor before and after FMT.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Hou, MD, Principal Investigator — Bejing Goboard Boren Hospital
Locations (1):
- Bejing Goboard Boren Hospital, Beijing, China